CLINICAL TRIAL: NCT05049681
Title: Anti-PD-1 Antibody SHR-1210 Combined With Apatinib Versus SHR-1210 in the Second-line Treatment of Advanced Esophageal Squamous Cell Carcinoma：A Multicentre，Randomized， Open Label，Phase 3 Study
Brief Title: Study of Anti-PD-1 Antibody SHR-1210 Plus Apatinib vs SHR-1210 as Second-Line Treatment of Advanced Esophageal Squamous Cell
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Feng Wang (Other)
Responsible Party: Sponsor-Investigator, Feng Wang, doctor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-EC020
Record Dates: First submitted 2021-09-13; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210（Camrelizumab）+Apatinib (Experimental): Apatinib 250mg, q.d.po; SHR-1210（Camrelizumab） 200 mg，Intravenous injection,q2W ,A course of treatment need 28 days.
  Interventions: Drug: Camrelizumab; Drug: Apatinib
- SHR-1210（Camrelizumab） (Active Comparator): SHR-1210（Camrelizumab） 200 mg，Intravenous injection. q2W ,A course of treatment need 28 days.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — SHR-1210（Camrelizumab） 200 mg，Intravenous injection， q2W ，A course of treatment need 28 days.
  Other Names: SHR-1210
Drug: Apatinib — Apatinib 250mg, q.d.po
  Arms: SHR-1210（Camrelizumab）+Apatinib

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of Anti-PD-1 antibody SHR-1210 plus apatinib versus SHR-1210 as second-line treatment of advanced esophageal squamous cell.

DETAILED DESCRIPTION:
The incidence of esophageal cancer is ranked seventh in the world, and the mortality rate ranks sixth in the world. At present, the first-line treatment of advanced esophageal cancer is mainly based on the combination of paclitaxel, cisplatin and fluorouracil. After the failure of first-line treatment, there is no standard second-line treatment. Recently the study of KEYNOTE181, ATTRACTION-3 and ESCORT had confirmed that PD-1 single drug in the second-line treatment of esophageal cancer is better than the previous traditional chemotherapy, and has become a new standard treatment. In order to further improve the therapeutic efficacy and prognosis of advanced esophageal squamous cell carcinoma, we designed this phase III clinical study to compare the efficacy and safety of shr-1210 combined with apatinib and shr-1210 in the second-line treatment of esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, males or females;
2. Histologically or cytologically confirmed as ESCC, locally advanced and unresectable, with local recurrence (local lymph node metastases) or distant metastases;
3. Having progressed or being intolerant to first-line systemic chemotherapy (including chemotherapy based on cisplatin, taxol or fluorouracil). Patients are also eligible if they progress after maintenance treatment following the first-line chemotherapy, or if patients with postoperative recurrence or metastasis progress after concurrent radiochemotherapy. As for the radical concurrent chemoradiotherapy, neoadjuvant/adjuvant treatment (chemotherapy or radiochemotherapy), if patients progress during the treatment or within six months after treatment, it is considered as a failure of first-line treatment;
4. According to the Response Evaluation Criteria In Solid Tumour (RECIST 1.1), there is at least one measurable lesion, which has not received any local treatment, such as radiotherapy (if the lesion within the region of the previous radiotherapy is confirmed to progress and satisfies RECIST1.1, it can be also selected as the target lesion) ;
5. Tissue samples should be provided for biomarker analysis. The newly harvested tissues are preferred. If the newly harvested tissues are not available, 5-8 archival paraffin sections (5 um thick) can be provided;
6. ECOG: 0~1;
7. Expected survival time ≥ 12 weeks;
8. Adequate function of major organs defined as:(1) Routine blood test: a. HB ≥ 90 g/L; b. ANC ≥ 1.5 × 109/L; c. PLT ≥ 80 × 109/L;(2) Biochemical test: a. ALB ≥ 30 g/L; b. ALT and AST ≤ 2.5 ULN; if there is no liver metastasis, ALT and AST ≤ 5 ULN; c. TBIL ≤ 1.5ULN; d. Plasma Cr ≤ 1.5 ULN or creatinine clearance rate (CCr) ≥ 60 mL/min;
9. Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
10. Women of childbearing age should consent to take contraception measures during the study period and within 6 months after the end of the study (eg., intrauterine device, oral contraceptive pills or condoms). The subjects must be negative for the serum or urine pregnancy test within 7 days before the recruitment. The female subjects must be non-lactating women. Males should consent to take contraception measures during the study period and within 6 months after the end of the study;
11. All subjects are recruited on a voluntary basis and sign the informed consent. They are required to be compliant with the study and cooperative with the follow-up.

Exclusion Criteria:

1. Patients who have any active autoimmune diseases or a past history of autoimmune diseases (including but not limited to the following: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, and hyperthyroidism; leukoderma. Subjects with fully remitted childhood asthma and no need for any intervention during adulthood can be included; those still having the need for bronchodilators for medical intervention cannot be included);
2. Patients who are currently on immunosuppressors or systemic hormone therapy for immunosuppressive purposes (dose > 10 mg/day, prednisone or other hormones with equivalent efficacy), and continue taking them within 2 weeks before recruitment;
3. ESCC patients with active bleeding in primary lesions;
4. ESCC patients in whom the primary lesions are not surgically resected and are not shrunken in size after radiotherapy;
5. Patients who have received treatment with VEGFR inhibitors, such as sorafenib, sunitinib, and apatinib;
6. Any of the following conditions that will interfere with oral medications: unable to swallow, having received gastroenterectomy, chronic diarrhea and intestinal obstruction;
7. Brain metastasis or brain metastases that have disappeared in less than 3 months;
8. Patients who have any severe and/or uncontrolled diseases, including: poor blood pressure control (systolic pressure ≥ 150 mmHg or diastolic pressure ≥ 100 mmHg); having myocardial ischemia or myocardial infarction and arrhythmia of Grade 1 and above (including QT interval ≥ 480 ms) and cardiac insufficiency of Grade 1; active or uncontrollable severe infection; liver diseases, such as decompensated liver failure, active hepatitis B (HBV-DNA ≥ 104 copy number/mL or 2000 IU/mL) or hepatitis C (positive for anti-HCV antibodies, and HCV-RNA higher than the lower limit of detection with the analytical method); routine urine test indicates urine protein ≥++ and confirms that the 24-hour urinary protein quantification>1.0 g;
9. Patients whose wounds or bone fractures remain unhealed for a long period of time;
10. Pneumorrhagia > NCI-CTC AE Grade1 within four weeks before recruitment; bleeding at other positions >NCI-CTC AE Grade 2 within four weeks before recruitment; having a bleeding tendency (eg., active peptic ulcer) or currently receiving thrombolytic or anticoagulant therapy, such as warfarin, heparin, or their analogs;
11. Patients who have experienced arterial/venous thrombotic events within six months, such as cerebrovascular accidents (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
12. The invasion of important blood vessels by the tumour or a high probability of the invasion of important blood vessels by the tumor that may lead to lethal hemorrhage in the study period ahead, as judged by the investigator according to the radiological examination;
13. Pregnancy or lactation;
14. Patients who have a history of other malignancies in the past five years (except for the cured basal cell carcinoma and cervical carcinoma in situ);
15. Patients who have a history of psychotropic drug abuse and unable to quit or having mental disorders;
16. Patients who have participated in other clinical trials of drugs in the past four weeks;
17. Patients who have concomitant diseases that may severely impair the safety of patients or make the patients unable to complete the study, as judged by the investigator;
18. Other patients who are considered inappropriate for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-12-05 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | up to 2 year
  the time from Randomization until death from any reason

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  the time from Randomization to the first disease progression or death from any cause
Objective Response Rate (ORR) | up to 1 year
  the proportion of patients with complete response or partial response determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Disease Control Rate (DCR) | up to 1 year
  the proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD)
Duration of response（DOR） | up to 2 year
  the time from the first response date to the first disease progression or death date
Time to response（TTP） | up to 1 year
  the time from treatment to first confirmed tumour response
6-, 9- and 12-month OS rates | up to 1 year
  overall survival rates at 6-, 9- and 12-month
adverse events(Safety) | up to 2 year
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University